CLINICAL TRIAL: NCT06627491
Title: Does the Speed of Imagined Muscle Contractions Affect Muscle Function and Central Nervous System Excitability?
Brief Title: Influence of Fast and Slow Imagined Muscle Contractions on Muscle Function or Central Nervous System Properties
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kennesaw State University (Other)
Responsible Party: Principal Investigator, Garrett Hester, Associate Professor of Exercise Science, Kennesaw State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MI_KA
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: Muscle strength; Nervous System; Motor Imagery
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Participants will rest quietly with eyes closed during the control condition.
- Fast (Experimental): Participants will imagine 2 blocks of 25 fast muscle contractions separated by 30 sec
  Interventions: Behavioral: Imagined muscle contractions
- Slow (Experimental): Participants will imagine 2 blocks of 25 slow muscle contractions separated by 30 sec
  Interventions: Behavioral: Imagined muscle contractions

INTERVENTIONS:
Behavioral: Imagined muscle contractions — The intervention involved imagining, with no physical movement, of muscle contractions.
  Arms: Fast; Slow

SUMMARY:
The goal of this randomized clinical trial is to learn if imagining fast or slow muscle contractions causes different responses for nervous system excitability and muscle function in young, healthy males and females in. The main questions are:

Does imagining fast muscle contractions cause greater nervous system excitability compared to imagining slow muscle contractions?

Does imagining fast muscle contractions increase muscle function compared to imagining slow muscle contractions?

A control condition (rest) will be compared with two intervention conditions: imagining fast and imagining slow conditions, to determine if the fast and slow increase outcomes more than control and if fast has the greatest response.

Participants will:

* Attend 4 laboratory visits
* Perform 50 imagined contractions fast or slow, but with no physical movement
* Physical muscle contractions and non-invasive brain stimulation would be completed before and after each condition.

DETAILED DESCRIPTION:
Participants will complete 4 laboratory visits in a randomized order, including a familiarization session, a control condition, and 2 conditions involving imaginary muscle contractions. During visits involving imaginary muscle contractions, participants will complete 2 sets of 25 repetitions of either fast (i.e., less than 1 second to peak torque increase torque as fast as possible) or slow (i.e., 3 seconds to peak torque) isometric elbow flexions. Before and after each condition, single-pulse transcranial magnetic stimulation will be delivered to the primary motor cortex to measure the amplitude of motor-evoked potentials and the duration of the resulting silent periods in the bicep brachii to quantify changes in corticospinal excitability and inhibition, respectively. Rapid maximal voluntary isometric contractions will be used to measure changes in rate of torque development, peak torque, and rate of muscle activation.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 - 30
* Healthy (no medical conditions)
* If female, must be taking the same monophasic oral contraceptive for the past 6 months
* Have a body mass index between 18.5 - 30 kg/m2
* Have not performed structured cardiovascular or resistance exercise in past 3 years
* Be right-handed
* Not currently taking stimulants, antipsychotic, anxiety, or depression medications
* Have not suffered an upper extremity musculoskeletal injury within the past year

Exclusion Criteria:

* If transcranial magnetic stimulation (TMS) is not deemed appropriate depending on your responses to the TMS-specific questionnaire
* Being ambidextrous
* Although rare, you will be excluded if discernable muscle activation responses are not possible via TMS

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male and female
Enrollment: 18 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in rate of torque development as measured by newton-meters per second | Baseline, minute 20
  A measure of the capacity to increase muscle torque rapidly as determined by the slope of the torque-time curve
Change in nervous system excitability as measured by electromyographic waveform aplitude following motor cortex stimulation | Baseline, minute 20
  A measure of excitability for the corticospinal tract

SECONDARY OUTCOMES:
Change in isometric bicep strength as measured by newton-meters of torque | Baseline, minute 20
  Isometric strength of a muscle
Change in agonist muscle activation as measured by electromyography amplitude | Baseline, minute 20
  A measure of the capacity at which the muscle is activated by the nervous system
Change in antagonist co-activation as measured by electromyography amplitude | Baseline, minute 20
  A measure of the capacity at which the antagonist muscle is activated by the nervous system
Change in rate of agonist muscle activation as measured by electromyography amplitude | Baseline, minute 20
  A measure of how quickly the nervous system activates the muscle
Change in nervous system inhibition as measured by electromyographic waveform aplitude following motor cortex stimulation | Baseline, minute 20
  A measure of inhibition for the corticospinal tract

OTHER OUTCOMES:
Self-reported ability to imagine movements as measured by Movement Imagery Questionnaire-Revised as measured on a scale from 8 to 56 | Baseline
  Survey that estimates one's capacity to imagine movement. A higher score indicates better imagination.
Level of vividness for imagining the imagined contractions as measured by 7-point likert scale as measured from 1 to 7 | 20 minutes after baseline
  A 7-point likert scale is used to to determine how vivid one's imagination was for the conditions. A higher score indicates greater difficulty imagining the movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Kennesaw State University, Kennesaw, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Non-identifying IPD will be provided upon a reasonable request.
Time Frame: Beginning 3 months and ending 5 years after the publication of results